CLINICAL TRIAL: NCT01765062
Title: One Year Skeletal and Dental Arch Changes Following Rapid Maxillary Expansion Treatment in Children
Acronym: ERM
Status: Completed | Type: Observational
Sponsor: State University of Maringá (Other)
Responsible Party: Principal Investigator, André Barbisan de Souza, DDS, Kelly Regina Micheletti, DDS, State University of Maringá
Other Study IDs: KRM-300585
Record Dates: First submitted 2012-12-20; First posted 2013-01-10 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Cross-bite
Keywords: Rapid maxillary expansion; Cross bite; Haas appliance; Lateral cephalograms
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Before Rapid Maxillary Expansion: T0
- 3 months After Rapid Maxillary Expansion: T1
- One year After Rapid Maxillary Expansion: T2

SUMMARY:
Many author have exposed the rapid and slow expansion, the diversity of activation and containment protocols and the follow-up time, justify the need for more studies to evaluate the effects to the ERM for the long-term.

ELIGIBILITY:
Inclusion Criteria:

* cross-bite with maxillary atresia

Exclusion Criteria:

* patients had undergone orthodontic treatment or had a syndrome

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2008-07; Primary Completion 2008-09 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
changes in cephalometric variables | prior to rapid maxillary expansion (T0), after three months (T1) and after one year

SECONDARY OUTCOMES:
Dental casts | prior to rapid maxillary expansion (T0), after three months (T1) and after one year (T2).

CONTACTS AND LOCATIONS:
Overall Officials: Daniela G Garib, PHD, Principal Investigator — Universidade de São Paulo-USP-Faculdade de Odontologia de Bauru
Locations (1):
- Universidade Estadual de Maringa, Maringá, Paraná, Brazil